CLINICAL TRIAL: NCT04162548
Title: Reaching the Frail Elderly for the Management of Atrial Fibrillation
Acronym: REAFEL
Status: Completed | Type: Observational
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Helena DOMINGUEZ, MD, PhD, Associate Professor, University Hospital Bispebjerg and Frederiksberg
Other Study IDs: H-18052892
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Atrial Fibrillation
Keywords: frail; public health
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cardio-relay: "Cardio-relay" is a novel collaboration model between hospital-based specialists and primary care, to provide high-quality care to frail patients, relieving their burden to attend multiple hospital specialist visits.
  Using telemedicine, it is possible to make measurements where the patient is (at the family clinic at the patient's home). Data are available for all the involved. That is, primary the patient, the relatives and caregivers that the patient wishes help from and health professionals from the family clinics and the hospital. Thereby, the hospital-based specialist supports the family clinic with expert knowledge, the need for attending the hospital facilities reduced to focus on what is strictly needed as specialized provider. Ultimately, the patient can be reached for high-quality care, relieving the patient's burden to attend multiple hospital specialist visits.

SUMMARY:
The overall objective of the project is to develop a collaboration model between the patient, the patient's General Practitioner (GP) and the cardiologist at the hospital in a seamless collaborative model dubbed the "Cardio-relay model".

The specific purpose of the pilot project is to ease performing heart rhythm monitoring with focus on diagnosis and evaluation of atrial fibrillation (AF), for patients who have difficulties to attend repeated visits to the hospital-based outpatient clinic.

With available eHealth technologies the cardiologist can access data gathered at the patient's side to provide support to the GP for selecting patients with need for heart rhythm monitoring, plan further evaluations and guide therapeutic decisions. These patients can thereby receive support that without the burden of attending physical meetings at the cardiologist office. The investigators evaluate if the cardio-relay model allows to complete evaluation of frail patients compared to usual care and if patients experience are sufficiently confident accessing the cardiologist through the cardio-relay model.

DETAILED DESCRIPTION:
Hypothesis Our overall hypothesis is, that using the cardio-relay model it is possible to provide adequate treatment to frail patients that have difficulties to attend repeated visits at the hospital-based cardiologist office.

Our concrete hypothesis is that a larger number of frail patients reaches adequate treatment with the cardio-relay model compared with conventional treatment and the patient remains confident with the distant support by the cardiologist.

METHODS This is a pragmatic clinical trial that uses mixed methods in different stages of the project to test this hypothesis. Observational during the initial feasibility period, an open-label cluster-randomization trial and an iterative implementation period.

Phase 1 - Feasibility During this phase, a single GP clinic is used to establish the elements that permit to establish the cardio-relay model. Hence, a field study is required to initiate the study.

Subsequently, the first of such elements in the cardio-relay model is a text exchange initiated by the GP addressing a request to the cardiologist to assess the need for heart rhythm monitoring. This is a replacement of usual referral when the cardiologist is expected to plan an appointment for the patient In the cardiology outpatient clinic or reject the referral. In the cardio-relay model, through a text exchange. The GP may require further examinations and add eventual results available in the hospital electronic records from previous contacts. The GP, the cardiologist and the patient (welcoming help from relatives and carers) can then agree on need for heart rhythm monitoring. The GP has available compact Holter sensors, C3+, from Cortrium ApS and can immediately initiate recordings at their office or at the patient's home. The duration of the recording is 24 hours as standard, but can agreed to prolong or repeat between the GP, the cardiologist and the patient. C3+ has memory for continuous electrocardiogram recording and built-in accelerometer, for up to three weeks and battery capacity for one weeks. The finalized recordings can be uploaded to the cloud by the GP and the cardiologist provides the GP with a result of the recording and a proposal for treatment according to the findings or further evaluation, which continuous the dialogue across the sectors

Phase 2 - Cluster randomization trial The terms of patient confidentiality are identic to those for usual care as patient management aims at best clinical practice according to local guidelines and data are recorded in the existing medical records. Hence, analysis of the observations gathered during Phase 1 correspond to those of a quality control project, with no requirement to gather specific informed consent for this part. The project has been accepted by the Ethics Committee of the Capital region (H-18052892) and published in clinicaltrials.gov for extending usual clinical management with questionnaires and structured interviews with patients to assess the satisfaction of the novel management with the cardio-relay model, with emphasis on the patient's perspective.

To allow comparison of the novel collaborative model cardio-relay with usual care, there will be conducted a cluster-randomization trial. Firstly, other GP clinics will be recruited by personal visit at the clinics where the cardio-relay model is briefly introduced. GP clinics will be invited to participate from different regions, that is, Bispebjerg-Frederiksberg municipality and Holbæk municipality, four from each municipality. That is eight GP clinics in total. During a subsequent workshop, the participant GP clinics will be invited to a workshop where they will be informed on the project and discuss best pathways to achieve the goals of the project, based on the principle of the project, adapted to the local GP characteristics. Collaboration agreements will be signed with the participant GP clinics they will be allocated to cluster by Region and randomized to intervention or no intervention. All sites send an initial message to the clinics to discuss the wish of Holter monitoring. In the control group, the initial requirement for Holter monitoring will be handled according to usual care. In the intervention group, GP will receive advise to start a C3+ Holter or not, eventually after a dialogue to qualify indication for Holter monitoring, and receive a treatment and further evaluation proposal, as described in the feasibility phase.

Measurements of efficacy will be initiated after the first two patients are managed in each site, both according to the control group and according to the intervention group. That is, 16 patients in total in the run-in period. It is planned to evaluate the results of Phase 2 when the first 50 patients are included and followed for six months (that is 16 patients run-in and 34 randomized). Measurements for the 34 patients managed according to randomization. This is an estimate based on an expected optimization of the following primary endpoint:

• Completion of evaluation for definite or roll-out diagnosis within six weeks in 90% of patients included in the intervention arm compared to 70% within six weeks These estimates are based on the time from referral to clinical visit for treatment decision or completed rule-out evaluation time in current settings on 120 patients referred to Bispebjerg-Frederiksberg hospital for evaluation for atrial fibrillation in the period January-June 2019 (mean 58 days, CI 11.27). This will be recalculated when the results of Phase 1 are available.

Questionnaires and patient interviews Questionnaires include validated assessment tools: Euro Quality of Life-5 Domain (EQ-5D) READY concept-based, psychometrically sound, validated instrument, the Readiness and Enablement Index for Health Technology (READHY), based on the concept of eHealth literacy supplemented with relevant scales from other instruments assessing aspects of self-management and social support: the eHealth Literacy Questionnaire (eHLQ) the Health Education Impact Questionnaire (heiQ) and the Health Literacy Questionnaire (HLQ).

Measurements

For questionnaires:

All instruments are based on conceptual dimensions and are rated on a Likert-type scale from 1 (strongly disagree) to 4 (strongly agree). The overall svore of each dimension is calculated as the mean of the items constituting the dimension.

For interviews:

All transcribed interviews will be were coded and categorized inductively using manifest qualitative content analysis, Qualitative data from the patient interviews will be reported in accordance with COREQ guidelines. Recruitment of patients for interviews will be prospective, with a "purposive approach. Every patient who agrees to take part in the project will be classified as "frail" or "not frail" pursuant to the pre-defined criteria (Table 1). Continuous comparison methods will be used to identify the population which could benefit from the cardio-relay model.

Table 1. "Frail elderly" are aged ≥ 65 years and have at least one of the following impairments:

* Transportation: Need for help to get to hospital outpatient departments
* Personal care: Need for help in personal hygiene
* Walking impairment: Reduced ability to walk (takes more than 5 sec. for the patient to walk 5 metres)
* Weight loss: Unintentional weight loss within the past year
* Cognitive difficulties: dementia, memory problems, aphasia, etc.
* Social problems: due to alcohol abuse or other abuse, ethnic background, language, etc.

Phase 3 - Iterative adjustment It is expectable that, after initial use of the cardio-relay model in REAFEL in the prior phases, there will be unforeseen improvement possibilities that can be adjusted in an iterative manner in the different settings for each participating sites. After a 6 months period it is expected to draw a generalizable guide for managing patients with the cardio-relay model.

Reporting results of the entire trial will follow TIDieR checklist.

ELIGIBILITY:
Inclusion Criteria:

* "Frail elderly" are aged ≥ 65 years
* Non-frail adults (> 18 years old)

Exclusion Criteria:

* Not willingness to participate

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients referred from primary care to assess atrial fibrillation diagnosis and burden "Frail elderly" are aged ≥ 65 years and have at least one of the following impairments:
  * Transportation: Need for help to get to hospital outpatient departments
  * Personal care: Need for help in personal hygiene
  * Walking impairment: Reduced ability to walk (takes more than 5 sec. for the patient to walk 5 metres)
  * Weight loss: Unintentional weight loss within the past year
  * Cognitive difficulties: dementia, memory problems, aphasia, etc.
  * Social problems: due to alcohol abuse or other abuse, ethnic background, language, etc.
Sampling Method: Probability Sample
Enrollment: 344 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Time to diagnosis conclusion | six months follow-up
  Completion of evaluation for definite or rule-out diagnosis within six weeks in 90% of patients included in the intervention arm compared to 70% within six weeks

SECONDARY OUTCOMES:
Identification of population that benefits with the cardio-relay model | six months follow-up
  patient satisfaction measured with focused interviews

OTHER OUTCOMES:
Number of referrals | six months follow-up
  Explorative analysis on number of referrals to the cardiology outpatient clinic

CONTACTS AND LOCATIONS:
Overall Officials: Helena DOMINGUEZ, MD, PhD, Study Chair — Frederiksberg hospital
Locations (1):
- Cardiology department Y, Bispebjerg-Frederiksberg Hospital, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bavelloni A, Piazzi M, Raffini M, Faenza I, Blalock WL. Prohibitin 2: At a communications crossroads. IUBMB Life. 2015 Apr;67(4):239-54. doi: 10.1002/iub.1366. Epub 2015 Apr 21. PMID 25904163
- [Result] Kayser L, Karnoe A, Furstrand D, Batterham R, Christensen KB, Elsworth G, Osborne RH. A Multidimensional Tool Based on the eHealth Literacy Framework: Development and Initial Validity Testing of the eHealth Literacy Questionnaire (eHLQ). J Med Internet Res. 2018 Feb 12;20(2):e36. doi: 10.2196/jmir.8371. PMID 29434011
- [Result] Osborne RH, Elsworth GR, Whitfield K. The Health Education Impact Questionnaire (heiQ): an outcomes and evaluation measure for patient education and self-management interventions for people with chronic conditions. Patient Educ Couns. 2007 May;66(2):192-201. doi: 10.1016/j.pec.2006.12.002. Epub 2007 Feb 22. PMID 17320338
- [Result] Osborne RH, Batterham RW, Elsworth GR, Hawkins M, Buchbinder R. The grounded psychometric development and initial validation of the Health Literacy Questionnaire (HLQ). BMC Public Health. 2013 Jul 16;13:658. doi: 10.1186/1471-2458-13-658. PMID 23855504
- [Result] Barbour RS. Checklists for improving rigour in qualitative research: a case of the tail wagging the dog? BMJ. 2001 May 5;322(7294):1115-7. doi: 10.1136/bmj.322.7294.1115. No abstract available. PMID 11337448
- [Result] Schiotz ML, Host D, Frolich A. Involving patients with multimorbidity in service planning: perspectives on continuity and care coordination. J Comorb. 2016 Sep 16;6(2):95-102. doi: 10.15256/joc.2016.6.81. eCollection 2016. PMID 29090180
- [Result] Rutter D, Manley C, Weaver T, Crawford MJ, Fulop N. Patients or partners? Case studies of user involvement in the planning and delivery of adult mental health services in London. Soc Sci Med. 2004 May;58(10):1973-84. doi: 10.1016/S0277-9536(03)00401-5. PMID 15020013